CLINICAL TRIAL: NCT02841891
Title: A Prospective, Randomized, Controlled, Multicenter Clinical Study Comparing Standard Anastomosis Closure Technique to Standard Closure Techniques Plus Sylys® Surgical Sealant
Brief Title: A Clinical Study Comparing Standard Anastomosis Closure Technique to Standard Closure Techniques Plus Sylys® Surgical Sealant
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Resource Constraints
Sponsor: Cohera Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO-106-0129
Record Dates: First submitted 2016-07-18; First posted 2016-07-22 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Colorectal and Ileorectal Anastomosis; Colocolic and Ileocolic Anastomosis; Coloanal and Ileoanal Anastomosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Test (Experimental): Test group will receive Sylys® Surgical Sealant as an adjunct to standard closure of stapled anastomosis in colectomy procedure.
  Interventions: Device: Sylys® Surgical Sealant
- Control (Active Comparator): Control group will receive standard of care closure of stapled anastomosis in colectomy procedure without Sylys® Surgical Sealant.
  Interventions: Procedure: Stapled Anastomosis Colectomy Procedure

INTERVENTIONS:
Device: Sylys® Surgical Sealant — Standard Stapled Anastomosis Colectomy Procedure with the addition of Sylys® Surgical Sealant
  Arms: Test
Procedure: Stapled Anastomosis Colectomy Procedure — Standard Stapled Anastomosis Colectomy Procedure without the addition of Sylys® Surgical Sealant
  Arms: Control

SUMMARY:
The Cohera Sylys® Surgical Sealant study is a prospective, randomized, controlled, multicenter clinical study comparing standard anastomosis closure technique (Control) to standard closure technique plus Sylys® Surgical Sealant (Test) in patients undergoing a colectomy procedure with a stapled anastomosis.

ELIGIBILITY:
Inclusion Criteria:

* Be 22 years of age or older
* Be scheduled for a colectomy procedure with a stapled anastomosis
* At time of surgery, has a completed anastomosis that is able to be visualized and is accessible to allow for circumferential sealant application with minimal bowel manipulation (≥90%)
* Completed anastomosis must be at a location where a WCE can be performed to evaluate for a sub-clinical leak
* Agree to return for all follow-up evaluations and procedures specified in the protocol
* Understand and give informed consent

Exclusion Criteria:

* Albumin < 3 g/dL
* ASA score (American Society of Anesthesiologists) ≥ 4
* Neutropenia ≤ 800 cells/µl
* Pregnant at time of surgery
* Has AIDS (HIV positive not excluded)
* Has neutropenia (IBD and steroid use not excluded)
* Has a known blood clotting disorder requiring treatment
* Has any condition known to effect wound healing, such as collagen vascular disease
* Has known or suspected allergy or sensitivity to any test materials, reagents, or WCE contrast materials
* Has undergone chemotherapy within 4 weeks of the anastomosis procedure and/or radiation within 3 days of the anastomosis procedure
* Concurrently using fibrin sealants or other anastomosis care devices
* Emergency surgery for abdominal indications
* Has undergone a colectomy procedure in the previous two months
* Has an emergent infection related to a previous colectomy procedure
* Is scheduled to undergo a Hartmann's procedure
* Is scheduled to undergo trans-anal endoscopic microsurgery (TEM)
* Is scheduled to undergo procedure using omental wrapping
* Is participating in another medical device trial involving colectomy with anastomosis

First 20 subjects ONLY:

• Is diagnosed with high risk cancer as determined by preoperative clinical evidence or diagnostic imaging (if patient's cancer stage has been downstaged through treatment prior to baseline screening, subject is allowed to be included):

* Lymph Node Cancer Stage: N2
* Cancer Tumor Size: T4
* Circumferential resection margin: CRM+ (Positive)

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-07; Primary Completion 2018-08-13 (Actual); Study Completion 2018-08-13 (Actual)

PRIMARY OUTCOMES:
Safety of Sylys® Surgical Sealant: Number of Anastomosis-Related Complications | 26 Weeks
  Number of subjects with anastomosis-related complications

SECONDARY OUTCOMES:
Sealant Application Evaluation Questionnaire | At time of device application (during surgery)
  Questionnaire documenting the ability to apply the sealant adequately to the anastomosis
Reduction in Anastomotic Leaks | 26 Weeks
  Comparison of anastomotic leak rate across all subjects

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Southern Alabama, Mobile, Alabama
  - University of California Irvine, Orange, California
  - University of Colorado Denver, Denver, Colorado
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Tulane, New Orleans, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Stony Brook University Hospital, Stony Brook, New York
  - Duke University, Durham, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor Scott & White Research Institute, Dallas, Texas
  - Houston Methodist, Houston, Texas
  - Intermountain Healthcare, Ogden, Utah
  - Univeristy of Utah, Salt Lake City, Utah